CLINICAL TRIAL: NCT01700803
Title: Povidone Iodine 10% Versus 7.5% Hand Scrub and Cesarean Section Wound Infections: A Randomized Trial
Brief Title: Povidone Iodine and Cesarean Section Wound Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Principal Investigator, Assiut University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Betadine CS
Record Dates: First submitted 2012-10-03; First posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Wound Infections
Keywords: Betadine; Povidine Iodine; Hand scrubbing; Cesarean section wound infections; post cesarean section
MeSH Terms: conditions — Wound Infection | interventions — Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Povidone Iodine 10% (Experimental): Using Povidone Iodine 10% hand scrub before caesarian section
  Interventions: Drug: Povidone Iodine 10% vand cesarean section wound infections
- Povidone Iodine 7.5% hand scrub (Experimental): Using Povidone Iodine 7.5% hand scrub before caesarian section
  Interventions: Drug: Povidone Iodine 7.5% vand cesarean section wound infections

INTERVENTIONS:
Drug: Povidone Iodine 10% vand cesarean section wound infections
  Arms: Povidone Iodine 10%
Drug: Povidone Iodine 7.5% vand cesarean section wound infections
  Arms: Povidone Iodine 7.5% hand scrub

SUMMARY:
The aim of this randomized clinical trial is to compare the efficiency of hand scrubbing by Povidone-Iodine solution 10% over 7.5% concentration in decreasing post-cesarean section wound infections & compare side effects of both agents.

DETAILED DESCRIPTION:
For centuries, hand washing with soap and water has been considered the main approach for personal hygiene. In the community, hand hygiene has been known to prevent infectious diseases and to decrease the burden of disease. Currently, hand hygiene is considered the most important measure for preventing the spread of pathogens in health-care settings.

There are multiple agents used for surgical hand scrubbing as alcohol, chlorhexidine, iodine/iodophors, para-chloro-meta-xylenol & triclosan. Ideally, the optimum antiseptic used for scrub should have broad spectrum of activity, persistent effect & fast acting. Unfortunately most studies evaluating surgical scrub antiseptics have focused on measuring hand bacterial colony counts. No randomized clinical trials have evaluated the impact of surgical scrub choice on surgical site infection risk & proven its efficiency.

ELIGIBILITY:
Inclusion Criteria:

* elective caesarian section (CS)

Exclusion Criteria:

* diabetes,
* immuno-compromised patients

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3231 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The difference of incidence of surgical site infection between both groups | 4 month
  Determine the difference in incidence of surgical site infection between Povidone Iodine 10% versus 7.5% hand scrub

SECONDARY OUTCOMES:
The difference in the side effects between both groups e.g. dermatitis | 4 month
  Determine the difference in incidence of side effects between Povidone Iodine 10% versus 7.5% hand scrub

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt